CLINICAL TRIAL: NCT02590107
Title: The Effect of Oral Supplementation and Improved Nutritional Status on Hematopoietic Stem Cell Transplant Patients
Brief Title: Early Oral Supplementation in Improving Nutritional Status in Patients Undergoing Hematopoietic Stem Cell Transplant
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE6Z14; NCI-2015-00477 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CASE6Z14 (Other: Case Comprehensive Cancer Center); P30CA043703 (NIH)
Record Dates: First submitted 2015-10-27; First posted 2015-10-28 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Malignant Neoplasm
MeSH Terms: conditions — Neoplasms | interventions — Dietary Supplements; Diet Records

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive care (Boost Plus, Pro-Stat 101) (Experimental): Participants receive Boost Plus PO BID or Pro-Stat 101 PO BID beginning one week before scheduled HSCT and continuing until hospital discharge. If participants do not tolerate the Boost Plus or Pro-Stat, they receive a milkshake PO QD as an alternative.
  Interventions: Dietary Supplement: Boost Plus; Dietary Supplement: Pro-Stat 101; Dietary Supplement: Milkshake; Other: daily food diaries

INTERVENTIONS:
Dietary Supplement: Boost Plus — Receive nutritional supplementation twice daily to provide 28g of protein
  Other Names: Supplementation
Dietary Supplement: Pro-Stat 101 — Receive nutritional supplementation twice daily to provide 30g of protein
  Other Names: Supplementation
Dietary Supplement: Milkshake — Receive alternate nutritional supplementation once daily to provide 28g protein
  Other Names: Supplementation
Other: daily food diaries — Participants will be given a food intake form, clipboard, and pen to record specific foods, as well as amounts of foods that are consumed from outside sources. In addition, the specific food items that each participant consumes will be recorded by the participant on his or her meal tickets which are included with each meal tray
  Other Names: food diary; food intake form

SUMMARY:
This clinical trial studies the use of early oral supplementation in improving nutritional status in participants undergoing hematopoietic stem cell transplant. Impaired nutritional status in participants undergoing hematopoietic stem cell transplant has been linked to decreased outcomes such as increased length of hospital stay and increased time to engraftment (an important milestone in transplant recovery). Early oral supplementation may increase nutritional status and help to promote a positive outcome in participants undergoing transplant.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if early oral supplementation improves nutritional status, decreases length of hospital stay, and shortens time to engraftment of hematopoietic stem cell transplant (HSCT) participants.

SECONDARY OBJECTIVES:

I. Serum albumin, serum 25-hydroxy vitamin D, and the degree of mucositis, as scored by the National Cancer Institute's Common Toxicity Criteria (NCI-CTC), a validated and widely accepted scale used for rating mucositis. The purpose of our secondary aims is to observe a potential correlation between the retrospective and prospective groups, as well as assess the need for future research based on these correlations.

OUTLINE:

Participants receive Boost Plus orally (PO) twice daily (BID) or Pro-Stat 101 PO BID beginning one week before scheduled HSCT and continuing until hospital discharge. If participants do not tolerate the Boost Plus or Pro-Stat, they receive a milkshake PO once daily (QD) as an alternative.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing an autologous or reduced intensity conditioning (RIC) allogeneic HSCT
* A serum albumin greater than or equal to 2.5 g/dL
* Able to understand and sign consent

Exclusion Criteria:

* Patients who have malabsorption problems, such as ulcerative colitis, irritable bowel syndrome, Crohn's disease, bowel surgery such as gastric bypass, and celiac disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Change in nutritional status determined by the Patient-Generated Subjective Global Assessment (PG-SGA) | Baseline to time of hospital discharge, up to 1 year
  To test the improvement of nutritional status over a period of time, a linear mixed model will be fit and the PG-SGA trend will be tested.

SECONDARY OUTCOMES:
Length of hospital stay, defined by time of admission through discharge | Up to time of hospital discharge, up to 1 year
  Longitudinal analysis of these ancillary variables will be performed to see the benefit of oral supplementation in the HSCT patients.
Change in serum albumin | Baseline, up to time of hospital discharge, up to 1 year
  Longitudinal analysis of these ancillary variables will be performed to see the benefit of oral supplementation in the HSCT patients.
Change in serum 25-hydroxy vitamin D | Baseline, up to time of hospital discharge, up to 1 year
  Longitudinal analysis of these ancillary variables will be performed to see the benefit of oral supplementation in the HSCT patients.
Degree of mucositis | Week 2, Week 3, Week 4, up to time of hospital discharge, up to 52 weeks
  Longitudinal analysis of these ancillary variables will be performed to see the benefit of oral supplementation in the HSCT patients.
Time to engraftment, defined by the first of three consecutive days that the absolute neutrophil count is greater than 500 | Up to time of hospital discharge, up to 1 year
  Longitudinal analysis of these ancillary variables will be performed to see the benefit of oral supplementation in the HSCT patients.

CONTACTS AND LOCATIONS:
Overall Officials: Autumn Diligente, MS, RDN, LD, Study Director — Case Comprehensive Cancer Center; Stephanie Logosh, MS, RDN, LD, Principal Investigator — Case Comprehensive Cancer Center
Locations (1):
- Case Comprehensive Cancer Center, Cleveland, Ohio, United States